CLINICAL TRIAL: NCT00341380
Title: Venous or Arterial Ligation and Intraoperative Dissemination (VALID) of Cancer Cells: A Randomized Clinical Trial For Patients With Resectable Non-Small Cell Lung Cancer
Brief Title: Prevention of Tumor Spread Due to Lung Cancer Surgery
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902319; 02-E-N319
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Cancer; Lung Cancer; Surgical Resection; Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients: Undergoing resection of lung tumor

SUMMARY:
This study will investigate operative techniques to reduce the risk of tumor spread as a result of lung cancer surgery. Recent studies indicate that tumor cells may be released into the bloodstream due to handling of the lung during surgery, causing disease spread in patients whose tumor was previously confined to the lung. This study will examine whether the order in which the pulmonary vein (a vessel carrying blood from the lungs to the heart) and artery (vessel carrying blood from the heart to the lungs) are tied off during surgery affects the risk of tumor spread and disease recurrence.

Patients 18 years of age or older with operable Stage I or Stage II non-small cell lung cancer and no evidence of tumor spread beyond the lung may be eligible for this study. Candidates will be screened with a medical history, blood tests, chest X-ray, and possibly mediastinal evaluation. This test involves inserting a tube into the chest cavity to look for signs of disease spread beyond the lung.

All participants will undergo standard surgery for lung cancer. During the procedure, both the pulmonary artery and pulmonary vein are tied off; for this study, patients will be randomly assigned to have either the artery or the vein ligated first. Patients will be followed every 6 months for two years with blood tests and X-rays to look for disease recurrence.

...

DETAILED DESCRIPTION:
The VALID study is designed to obtain information regarding factors associated with the risk of recurrence after resection of early stage Non-Small Cell Lung Cancer (NSCLC). Until recently, the only clearly identified prognostic factor was the stage of the disease. Recent development of sensitive molecular assays has provided a way to study the effect of circulating tumor cells on clinical outcome. Preliminary studies have shown that tumor cells detected by such means in lymph nodes or in bone marrow are associated with an increased risk of recurrence. Preliminary studies have also indicated that the level of circulating tumor cells in the blood stream is effected by intraoperative factors, i.e. the sequence of vessel ligation.

The main objective for this study is to investigate the influence of intraoperative sequence of vessel ligation and how this affects tumor recurrence and survival. In addition, we will also investigate the use of molecular assays to detect circulating tumor cells as a surrogate endpoint for the occurrence of distant metastases and/or death after surgery for NSCL. Several of these molecular markers have proven their value in case series but have not been rigorously tested for association with the clinical endpoints of interest, tumor recurrence and survival. We believe that this study may lead to important answers about how the spread of tumor cells occurs and if novel detection methods can be used to predict patient outcome.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients for this study will be identified through the Multidisciplinary Thoracic Oncology Clinic at UNC. Enrollment criteria for the study are: 1) Surgically respectable Stage I or II non-small cell lung carcinoma; 2) Negative mediastinal evaluation; 3) No contraindications for surgery; and 4) More than 18 years of age.

EXCLUSION CRITERIA:

Patients with prior carcinoma within 5 years (except basal cell carcinoma of the skin and superficial bladder cancer) will be excluded from the study. Patients who are enrolled based on clinical Stage I or II but are revised to higher Stage once the surgical specimens are examined will be excluded from statistical analysis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 or older with Stage I or II non-small cell lung cancer and no evidence of tumor spread beyond the lung.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2002-09-24; Primary Completion 2007-04-13 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Determine the effect of initial venous versus arterial ligation during resection for NSCLC on the risk of distant metastases within two years of follow-up | 2 years
  Risk of metastases recurrence after tumor resection

CONTACTS AND LOCATIONS:
Overall Officials: Jack Taylor, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Hansen E, Wolff N, Knuechel R, Ruschoff J, Hofstaedter F, Taeger K. Tumor cells in blood shed from the surgical field. Arch Surg. 1995 Apr;130(4):387-93. doi: 10.1001/archsurg.1995.01430040049007. PMID 7710337
- [Background] Kurusu Y, Yamashita J, Hayashi N, Mita S, Fujino N, Ogawa M. The sequence of vessel ligation affects tumor release into the circulation. J Thorac Cardiovasc Surg. 1998 Jul;116(1):107-13. doi: 10.1016/s0022-5223(98)70248-x. PMID 9671904
- [Background] Pantel K, Izbicki J, Passlick B, Angstwurm M, Haussinger K, Thetter O, Riethmuller G. Frequency and prognostic significance of isolated tumour cells in bone marrow of patients with non-small-cell lung cancer without overt metastases. Lancet. 1996 Mar 9;347(9002):649-53. doi: 10.1016/s0140-6736(96)91203-9. PMID 8596379